CLINICAL TRIAL: NCT02081911
Title: Postoperative Pain Management Following Total Knee Arthroplasty Utilizing Adductor Canal Block: Effects on Pain Management and Quadriceps Sparing
Brief Title: Total Knee Arthroplasty Utilizing Adductor Canal Block: Effect on Quadriceps Sparing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB #2014-005
Record Dates: First submitted 2014-02-28; First posted 2014-03-07 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Osteoarthritis (Knee)
Keywords: adductor canal; femoral; quadriceps
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- High volume Adductor canal block (Experimental): Adductor canal block performed in the distal thigh (1/3 of the total distance between the superior border of the patella and the femoral crease, cephalad to the patella) utilizing an injectate volume of 30 mL 0.25% bupivacaine/ epinephrine
  Interventions: Procedure: High Volume Adductor Canal Block
- Low volume Adductor Canal Block (Experimental): Adductor canal block performed in the distal thigh (1/3 of the total distance between the superior border of the patella and the femoral crease, cephalad to the patella) utilizing an injectate volume of of 10 mL 0.75% bupivacaine/ epinephrine
  Interventions: Procedure: Low Volume Adductor Canal Block
- Femoral nerve block (Experimental): Femoral nerve block with 10 mL 0.75 % bupivacaine/epinephrine
  Interventions: Procedure: Femoral Nerve Block

INTERVENTIONS:
Procedure: High Volume Adductor Canal Block — Adductor canal block performed in the distal thigh (1/3 of the total distance between the superior border of the patella and the femoral crease, cephalad to the patella) utilizing an injectate volume of 30 mL 0.25% bupivacaine/ epinephrine
  Arms: High volume Adductor canal block
Procedure: Low Volume Adductor Canal Block — Adductor canal block performed in the distal thigh (1/3 of the total distance between the superior border of the patella and the femoral crease, cephalad to the patella) utilizing an injectate volume of of 10 mL 0.75% bupivacaine/ epinephrine
  Arms: Low volume Adductor Canal Block
Procedure: Femoral Nerve Block — Femoral nerve block with 10 mL 0.75 % bupivacaine/epinephrine
  Arms: Femoral nerve block

SUMMARY:
The purpose of this study is to investigate whether there is quantitative motor-sparing of the quadriceps muscles following adductor canal nerve block versus femoral nerve block. Patients will be randomly placed into one of three treatment groups: 1) Femoral nerve block, 2) Adductor canal nerve block - low volume, or 3) Adductor canal nerve block - high volume. Quadriceps function will be assessed in the operating room using a skin patch and electrical stimulation. Follow up visits with the patients will continue over the course of 2 days during patient's stay at the hospital. A total of 60 patients will be enrolled for the study.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing primary unilateral total knee arthroplasty
* Planned use of combined spinal epidural (CSE) anesthesia
* Ability to follow study protocol

Exclusion Criteria:

* Contraindication to a spinal or epidural anesthetic
* Chronic opioid use (defined as daily or almost daily use of opioids for >3 months)
* Allergy to local anesthetics
* Pre-existing neuropathy or weakness of the operative limb
* Any neuromuscular disorder
* Diabetes type I and II
* Contraindication to a femoral nerve block or adductor canal nerve block
* Allergy or intolerance to any of the study medications
* BMI > 35 kg/m2

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Quadriceps function as assessed by non-invasive transcutaneous nerve stimulation of the femoral nerve | 15 minutes after the placement of the peripheral nerve block (femoral or adductor canal)
  After CSE effect, but prior to peripheral block, quadriceps function will be assessed by non-invasive transcutaneous nerve stimulation of the femoral nerve by placing an ECG electrode over the femoral location (determined by U/S) in the inguinal groove. The threshold amperage that produces patellar motion in response to electrical stimulation will be recorded. This threshold amperage will serve as a baseline value. Following the peripheral nerve block, transcutaneous stimulation will be repeated and, if still possible to elicit quadriceps contractions in response to electrical stimulation, the resulting new threshold amperage will be measured. The new threshold amperage will be expressed as a percentage of the baseline value and serve as a quantitative functional indication of the extent of quadriceps paresis resulting from the peripheral nerve block. The primary outcome will be quadriceps paralysis - yes/no.

SECONDARY OUTCOMES:
Threshold amperage as a percentage of the baseline value | 15 minutes after the placement of the peripheral nerve block
  Following the peripheral nerve block, transcutaneous stimulation will be repeated and, if still possible to elicit quadriceps contractions in response to electrical stimulation, the resulting new threshold amperage will be measured. The new threshold amperage will be expressed as a percentage of the baseline value and serve as a quantitative functional indication of the extent of quadriceps paresis resulting from the peripheral nerve block.
Analgesic adequacy | Resolution of the spinal anesthetic (2 hours post-op), 24 and 48 hours post-op
  Analgesic adequacy as determined by pain scores (0-10) at spinal resolution (on average 2 hours post-op), 24 hours post-op and 48 hours post-op and daily epidural patient controlled analgesia consumption
Ability to complete a straight leg lift | Holding area (baseline), at spinal resolution (2 hours post-op), 24 hours post-op and 48 hours post-op
  Ability to complete and hold (for 3 seconds) a straight leg lift (from supine position) against gravity as evidence of meaningful quadriceps function - performed in holding area (baseline), at spinal resolution (on average 2 hours post-op), 24 hours post-op and 48 hours post-op

CONTACTS AND LOCATIONS:
Overall Officials: William Urmey, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Result] Vloka JD, Hadzic A, Lesser JB, Kitain E, Geatz H, April EW, Thys DM. A common epineural sheath for the nerves in the popliteal fossa and its possible implications for sciatic nerve block. Anesth Analg. 1997 Feb;84(2):387-90. doi: 10.1097/00000539-199702000-00028. PMID 9024035
- [Result] Davis JJ, Bond TS, Swenson JD. Adductor canal block: more than just the saphenous nerve? Reg Anesth Pain Med. 2009 Nov-Dec;34(6):618-9. doi: 10.1097/AAP.0b013e3181bfbf00. No abstract available. PMID 19901788
- See also: Related Info — http://www.hss.edu